CLINICAL TRIAL: NCT07323290
Title: Twelve-Month Short-Term Marginal Bone Remodeling at Monolithic Zirconia Full-Arch Prostheses in the Maxilla and Mandible: A Clinical Study
Brief Title: Marginal Bone Remodeling at Monolithic Zirconia Full-Arch Prostheses in the Maxilla and Mandible
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Luis Carlos Garza Garza, Professor of Restorative Dentistry, Universitat Internacional de Catalunya
Other Study IDs: REST-ECL-202002
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Edentulism; Implant Dentistry
Keywords: Monolithic zirconia; V-shaped mandible; U-shaped mandible; Mandibular morphology; Bone remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maxilla group: 25 full-arch zirconia prostheses
  Interventions: Other: No intervention
- Mandible group: 24 full-arch zirconia prostheses
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. No experimental intervention is assigned. All treatments were performed as part of routine clinical care.

SUMMARY:
This prospective observational clinical study aims to compare 12-month clinical, radiographic, and patient-reported outcomes of monolithic zirconia full-arch implant-supported prostheses placed in the maxilla versus the mandible. The study also investigates whether mandibular morphology (U-shaped vs V-shaped) and arch geometry (inter-implant distance and cantilever length) are associated with early marginal bone remodeling. All arches were rehabilitated following standardized surgical and digital prosthetic protocols.

DETAILED DESCRIPTION:
This prospective observational cohort study investigates early marginal bone remodeling in full-arch implant-supported monolithic zirconia prostheses placed in the maxilla and mandible. Although monolithic zirconia has become a widely adopted restorative material due to its mechanical strength, esthetic stability, and reduced risk of veneering complications, limited evidence exists regarding whether early bone remodeling differs between the maxillary and mandibular arches or whether mandibular anatomical configurations influence these remodeling patterns. The present study was designed to address these knowledge gaps under rigorously standardized surgical and prosthetic conditions.

All participants were fully edentulous and rehabilitated following identical clinical protocols. Each arch received between six and eight titanium implants placed through computer-guided surgery, followed by the connection of multi-unit abutments and the delivery of an immediate-loading PMMA provisional prosthesis within 48 hours. After a healing period of three months, definitive monolithic zirconia full-arch prostheses were fabricated and delivered using a fully digital workflow. Standardized periapical radiographs were obtained at baseline (prosthesis insertion) and at the 12-month follow-up using customized positioning devices, fixed exposure parameters, and a paralleling technique to ensure reproducibility. Radiographs were calibrated digitally using the known implant thread pitch, and marginal bone level changes were measured by two independent calibrated examiners.

A key component of this study is the incorporation of mandibular anatomical variability into the analysis. Mandibular morphology was categorized into U-shaped and V-shaped configurations according to validated CBCT criteria based on intercanine-to-intermolar width ratios and anterior arch angles. Because mandibular flexure and strain distribution have been hypothesized to vary according to arch shape, the study evaluates whether these morphological classifications correspond to differences in early marginal bone remodeling. Additionally, geometric variables-including inter-implant distance and distal cantilever length-were extracted directly from the definitive CAD designs to assess potential associations between implant distribution and remodeling outcomes.

The study also incorporates patient-reported outcomes to better understand the functional and psychosocial impact of treatment. The OHIP-14 questionnaire and a visual analog scale (VAS) for satisfaction were administered at baseline and at the 12-month recall appointment. Clinical parameters, prosthetic complications, and peri-implant soft-tissue conditions were documented to complement the radiographic evaluation.

This design allows for multiple levels of comparison:

* Arch-level comparison (maxilla vs mandible) under identical surgical/prosthetic protocols.
* Morphology-specific analysis within the mandible (U-shaped vs V-shaped).
* Geometry-based evaluation assessing correlations between implant positioning (inter-implant distance, cantilever length) and marginal bone remodeling.
* Within-subject comparison for individuals rehabilitated in both arches.

Because the study is observational and non-interventional, it does not assign treatments or modify clinical protocols. Instead, it seeks to characterize natural remodeling patterns under contemporary full-arch zirconia rehabilitation techniques and to explore whether anatomical and geometric factors contribute to variability in early outcomes.

The broader goal of this research is to clarify whether certain mandibular anatomical configurations may benefit from modified implant distribution, segmented framework designs, or alternative prosthetic considerations. The findings have the potential to inform future guidelines in digital full-arch implant rehabilitation and help clinicians better anticipate patient-specific biomechanical challenges. Long-term follow-up and biomechanical measurements are encouraged for future studies to validate the associations observed in this 12-month analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 50 years old
* Edentulous maxilla or mandible
* Sufficient bone volume for implant placement
* Non-smokers or light smokers (<10 cigarettes/day)
* Able to provide informed consent

Exclusion Criteria:

* Bruxism
* Uncontrolled systemic diseases
* Bisphosphonate therapy
* Contraindications to dental implant surgery
* Active oral pathology

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Edentulous adults undergoing full-arch rehabilitation with monolithic zirconia prostheses at the Universitat Internacional de Catalunya and associated private practice centers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Loss (mm) | Baseline and 12 months
  Marginal bone loss will be measured as the change in peri-implant marginal bone level (in millimeters) between baseline (prosthesis delivery) and the 12-month follow-up. Measurements will be obtained from standardized periapical radiographs using a paralleling technique and calibrated based on implant thread pitch.
  Higher values indicate greater bone loss (worse outcome).

SECONDARY OUTCOMES:
Implant and Prosthetic Survival Rate | Baseline to 12 months
  Survival rate will be defined as the percentage of implants and prostheses remaining functional without loss, fracture, removal, or need for replacement.
  An implant or prosthesis is considered a failure if it requires removal, becomes fractured, or cannot maintain clinical function.
  Higher percentages indicate better survival outcomes.
Patient-Reported Outcomes (OHIP-14) | Baseline and 12 months
  Patient-reported oral health-related quality of life will be assessed using the OHIP-14 questionnaire, scored from 0 to 56, where:
  Higher scores indicate worse quality of life.
Patient-Reported Outcomes (Visual Analog Scale) | Baseline and 12 months
  Satisfaction will be measured using a Visual Analog Scale (VAS) from 0 to 10, where:
  0 = Not satisfied at all
  10 = Extremely satisfied
  Higher scores indicate greater satisfaction.
  Changes between baseline and 12 months will be reported.
Mechanical and Biological Complications | Baseline to 12 months
  Complications will include mechanical events (e.g., chipping, framework fracture, screw loosening) and biological events (e.g., soft-tissue inflammation, infection).
  Each event will be recorded as present (yes/no) and categorized according to type.
  Higher counts indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Roig, Phd, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Universitat internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
All data will be published

REFERENCES:
- [Background] Sivaraman K, Chopra A, Venkatesh SB. Clinical importance of median mandibular flexure in oral rehabilitation: a review. J Oral Rehabil. 2016 Mar;43(3):215-25. doi: 10.1111/joor.12361. Epub 2015 Oct 25. PMID 26498998
- [Background] Riera C, Karasan D, Sailer I, Mojon P, Fehmer V, Pitta J. Mechanical stability of posterior implant-supported monolithic zirconia cantilever on titanium-base abutments. An in vitro study. Clin Oral Implants Res. 2024 Aug;35(8):1042-1053. doi: 10.1111/clr.14251. Epub 2024 Feb 28. PMID 38415804
- [Background] Waltenberger L, Bishti S, Wolfart S. German S3 guideline on implant-supported all-ceramic restorations. Int J Implant Dent. 2025 Aug 13;11(1):53. doi: 10.1186/s40729-025-00641-7. PMID 40802222
- [Background] Todaro C, Cerri M, Rodriguez Y Baena R, Lupi SM. Lower Jaw Full-Arch Restoration: A Completely Digital Approach to Immediate Load. Healthcare (Basel). 2024 Jan 28;12(3):332. doi: 10.3390/healthcare12030332. PMID 38338217
- [Background] Garza LC, Crooke E, Valles M, Soliva J, Rodriguez X, Rodeja M, Roig M. Evaluation of Polymethyl Methacrylate as a Provisional Material in a Fully Digital Workflow for Immediate-Load Complete-Arch Implant-Supported Prostheses over Three Months. Materials (Basel). 2025 Jan 26;18(3):562. doi: 10.3390/ma18030562. PMID 39942227

DOCUMENTS (2):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT07323290/Prot_000.pdf
  • Informed Consent Form (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT07323290/ICF_001.pdf